CLINICAL TRIAL: NCT02189564
Title: Die Auswirkung Von Dopaminergen Belohnungsreizen Auf Das Lernen Einer Motorischen Fertikgeit Bei Gesunden Probanden "Effects of Dopaminergic Reward on Motor Skill Learning in Healthy Subjects"
Brief Title: Rewarding Feedback in Motor Learning and Rehabilitation
Acronym: KFSP-REWARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kai Lutz, PhD (Industry)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Kai Lutz, PhD, Scientific Director, Cereneo AG
Organization: Cereneo AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KFSP-SUB1-LU13054
Record Dates: First submitted 2014-06-30; First posted 2014-07-14 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Motor Performance; Motor Learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intrinsic reward (Active Comparator): Feedback about good performance
  Interventions: Behavioral: Feedback about good performance
- Intrinsic and extrinsic reward (Experimental): Feedback about good performance + money
  Interventions: Behavioral: Feedback about good performance + money
- Intrinsic reward (average performance) (Experimental): Feedback about random selection of trials
  Interventions: Behavioral: Feedback about average performance

INTERVENTIONS:
Behavioral: Feedback about good performance
  Arms: Intrinsic reward
Behavioral: Feedback about good performance + money
  Arms: Intrinsic and extrinsic reward
Behavioral: Feedback about average performance
  Arms: Intrinsic reward (average performance)

SUMMARY:
The effect of rewarding vs. non-rewarding feedback on acquisition of a motor skill is investigated in a single blinded parallel group design. Reward consists of performance dependent monetary reward, or of knowledge of performance in selected (above average) trials.

The investigators hypothesize improved motor skill learning and higher involvement of the dopaminsrgic system under rewarding vs. non-rewarding conditions.

ELIGIBILITY:
Inclusion Criteria:

* neurologically healthy
* right handed

Exclusion Criteria:

* Contraindications against magnetic resonance imaging
* pregnancy

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Motor skill learning using an arc pointing task | about 10 minutes pre-training, about 10 min post training, about 24h post training
  temporal and spacial precision in an arc pointing task will be assessed using 5 different movement speeds during the above mentioned time periods before and after a specific motor learning programm. Learning will be assessed as change from pre-training to post training

CONTACTS AND LOCATIONS:
Locations (1):
- Cereneo, Center For Rehabilitation and Neurology, Vitznau, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Widmer M, Ziegler N, Held J, Luft A, Lutz K. Rewarding feedback promotes motor skill consolidation via striatal activity. Prog Brain Res. 2016;229:303-323. doi: 10.1016/bs.pbr.2016.05.006. Epub 2016 Jul 7. PMID 27926445